CLINICAL TRIAL: NCT06706830
Title: The Role of Lung and Diaphragm Ultrasonography in Predicting Clinical Progression in Patients Receiving High-Flow Nasal Oxygen and Non-Invasive Mechanical Ventilation Support for Hypoxemic Respiratory Failure
Brief Title: The Role of Lung and Diaphragm Ultrasonography in Predicting Clinical Progression in Hypoxemic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Simge Evren (Other)
Responsible Party: Sponsor-Investigator, Simge Evren, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: 291
Record Dates: First submitted 2024-11-11; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Diaphragm Ultrasonography; Lung Ultrasound; Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hypoxemic: Patients whose partial oxygen levels are low

SUMMARY:
The goal of this observational study is to evaluate whether the risk of intubation in patients with hypoxemic respiratory failure who were monitored in the intensive care unit and received non-invasive mechanical ventilation and high-flow nasal oxygen treatment could be predicted using lung and diaphragm ultrasound.

The main question it aims to answer is:

Can lung and diaphragm ultrasound predict the risk of intubation in patients with hypoxemic respiratory failure?

DETAILED DESCRIPTION:
Between January 1, 2024, and May 1, 2024, the diaphragm thickness fraction, excursion, LUS score, ROX index, and the LUSS/ROX index ratio were evaluated using lung and diaphragm ultrasound in 91 patients admitted to the intensive care unit with a diagnosis of hypoxemic respiratory failure. These evaluations were performed at the 6th, 12th, 24th, and 48th hours of their ICU stay, and during intubation if the decision for intubation was made

ELIGIBILITY:
Inclusion Criteria:

-PaO2 <60 mmHg detected in arterial blood gas samples at the time of admission to the intensive care unit

Exclusion Criteria:

* Under the age of 18
* History of lung and diaphragm surgery
* Congenital, acquired or traumatic diaphragmatic hernia
* Diaphragm paralysis
* Hemodynamic instability requiring vasoactive drug support
* Do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypoxemic patients in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Lung and diaphragm ultrasound evaluation for risk of intubation | 48 hours
  Lung and diaphragm ultrasound can predict risk of intubation

SECONDARY OUTCOMES:
ROX index evaluation for risk of intubation | 48 hours
  The Respiratory Rate-Oxygenation Index can predict the risk of intubation Higher score means lower risk
LUSS/ROX index ratio evaluation for risk of intubation | 48 hours
  LUSS/ROX index ratio can predict the risk of intubation

CONTACTS AND LOCATIONS:
Overall Officials: Namigar Turgut, Study Director — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (2):
- Turkey (Türkiye) (2):
  - Prof. Dr. Cemil Tascıoglu City Hospital, Istanbul, Şişli
  - Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization, Istanbul, Şişli